CLINICAL TRIAL: NCT01714479
Title: Skeletal Muscle and Physical Performance Responses to Leucine-Enriched Nutrition Supplementation During Load Carriage
Brief Title: Skeletal Muscle Response to Amino Acids and Load Carriage Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: US Army Natick Soldier Research, Development & Engineering Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 12-18-HC
Record Dates: First submitted 2012-10-23; First posted 2012-10-26 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2016-09

CONDITIONS: Muscle Loss; Muscle Anabolism; Muscle Performance
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Load Carriage - Control (Placebo Comparator): Load Carriage - with a calorie-free placebo
  Interventions: Other: Placebo
- Load Carriage - leucine-enriched nutrition supplement (Experimental): Load Carriage with leucine-enriched amino acid supplementation
  Interventions: Other: Leucine-enriched nutritional supplement
- Conventional Exercise - Control (Placebo Comparator): Conventional Exercise with a calorie-free placebo
  Interventions: Other: Placebo
- Conventional Exercise - Leucine-enriched Nutrition Supplement (Active Comparator): Conventional Exercise with leucine-enriched Amino Acid supplementation
  Interventions: Other: Leucine-enriched nutritional supplement

INTERVENTIONS:
Other: Leucine-enriched nutritional supplement — A protein and carbohydrate supplement with high levels of leucine
  Arms: Conventional Exercise - Leucine-enriched Nutrition Supplement; Load Carriage - leucine-enriched nutrition supplement
Other: Placebo
  Arms: Conventional Exercise - Control; Load Carriage - Control

SUMMARY:
Warfighters often experience physical overload, as the uniform and associated gear that they carry burdens them with substantial loads. The loads increase energy expenditure to levels that exceed a Warfighter's typical energy intake. The typical assault load is approximately 25 kg, although loads as high as 55 kg are often carried, which when combined with extreme energy expenditures can degrade health and performance, and increase the risk of injury. Branched-chain amino acid (leucine) supplementation may confer protection against the negative effects of operational stress by stimulating muscle protein synthesis and reducing degradation. This study will determine if leucine-enriched nutrition supplementation confers protection against the negative consequences of sustained load carriage exercise, and explore the mechanisms by which leucine might impart protection.

ELIGIBILITY:
Inclusion Criteria:

* Weight stable (±5 lbs)with a body mass index between 22-29 kg/m2 and a VO2peak of 40 - 60 ml/kg/min
* Willing to refrain from taking any NSAIDS (i.e., aspirin, Advil®, Aleve®, Naprosyn®), or any aspirin-containing products, alchohol, and nicotine
* Females must be on oral contraception

Exclusion Criteria:

* Metabolic or cardiovascular abnormalities, gastrointestinal disorders
* Disease or medication that affects macronutrient metabolism or the ability to participate in strenuous exercise
* Allergies or intolerance to foods (e.g. lactose intolerance/milk allergy), vegetarian practices, or medications (including, but not limited to, lidocaine or phenylalanine) to be used in the study
* Anemia (HCT <38) and Sickle Cell Anemia/Trait, abnormal PT/PTT test or problems with blood clotting
* Present condition of alcoholism, use of nutritional/sports supplements, anabolic steroids, or other substance abuse issues
* Musculoskeletal injuries that compromise the ability to exercise
* Blood donation within 8 weeks of enrollment
* Pregnancy and women not on oral contraceptives

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in muscle protein synthesis and whole-body protein turnover during and after load carriage or conventional exercise with or without amino acid supplementation | 90 min exercise bout (exercise) and 180 min of recovery

SECONDARY OUTCOMES:
Changes in muscle performance in recovery from load carriage or conventional exercise with or without amino acid supplementation | 4, 24, 48, and 72 hours post exercise

CONTACTS AND LOCATIONS:
Overall Officials: Stefan M Pasiakos, Ph.D., Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Margolis LM, McClung HL, Murphy NE, Carrigan CT, Pasiakos SM. Skeletal Muscle myomiR Are Differentially Expressed by Endurance Exercise Mode and Combined Essential Amino Acid and Carbohydrate Supplementation. Front Physiol. 2017 Mar 23;8:182. doi: 10.3389/fphys.2017.00182. eCollection 2017. PMID 28386239
- [Result] Pasiakos SM, McClung HL, Margolis LM, Murphy NE, Lin GG, Hydren JR, Young AJ. Human Muscle Protein Synthetic Responses during Weight-Bearing and Non-Weight-Bearing Exercise: A Comparative Study of Exercise Modes and Recovery Nutrition. PLoS One. 2015 Oct 16;10(10):e0140863. doi: 10.1371/journal.pone.0140863. eCollection 2015. PMID 26474292
- [Derived] Margolis LM, Murphy NE, Carrigan CT, McClung HL, Pasiakos SM. Ingesting a Combined Carbohydrate and Essential Amino Acid Supplement Compared to a Non-Nutritive Placebo Blunts Mitochondrial Biogenesis-Related Gene Expression after Aerobic Exercise. Curr Dev Nutr. 2017 May 23;1(6):e000893. doi: 10.3945/cdn.117.000893. eCollection 2017 Jun. PMID 29955707